CLINICAL TRIAL: NCT07359274
Title: Clinical and Morphological Effects of Neurodynamic Mobilization and Carpal Bone Mobilization Techniques in Patients With Mild-to-Moderate Carpal Tunnel Syndrome
Brief Title: Effects of Neurodynamic and Carpal Bone Mobilization in Mild-to-Moderate Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Merve Akdeniz Leblebicier, Assoc. Prof., Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurodynamic and Carpal Mobs
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome; Splints
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neurodynamic mobs in addition splint (Experimental): Median nerve neurodynamic mobilization exercises administered by a physiotherapist for 4 weeks in addition to night-time wrist splint use
  Interventions: Other: Neurodynamic mobilization; Other: Splint
- Carpal Bone Mobilization + Splint (Experimental): Carpal bone mobilization techniques administered by a physiotherapist for 4 weeks in addition to night-time wrist splint use.
  Interventions: Other: Carpal bone mobilization; Other: Splint
- Splint only (Active Comparator): Neutral-position wrist splint worn at night for 4 weeks.
  Interventions: Other: Splint

INTERVENTIONS:
Other: Neurodynamic mobilization — Median nerve neurodynamic mobilization exercises performed 5 sessions per week for 4 weeks.
  Arms: neurodynamic mobs in addition splint
Other: Carpal bone mobilization — Manual carpal bone mobilization techniques applied 5 sessions per week for 4 weeks.
  Arms: Carpal Bone Mobilization + Splint
Other: Splint — Neutral-position wrist splint used during night-time for 4 weeks.

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy caused by compression of the median nerve at the wrist. Conservative interventions such as splinting and manual therapy are frequently used in individuals with mild-to-moderate CTS. Neurodynamic mobilization and carpal bone mobilization aim to improve neural and soft tissue mobility; however, their comparative effects on clinical outcomes and median nerve morphology are not fully understood.

This interventional, non-randomized clinical study aims to compare the clinical and ultrasonographic effects of neurodynamic mobilization plus splinting, carpal bone mobilization plus splinting, and splinting alone in patients with mild-to-moderate CTS. Ninety-three participants diagnosed with mild-to-moderate carpal tunnel syndrome based on electrodiagnostic criteria will be included. Participants will be allocated into three parallel groups without randomization. All participants will receive a neutral-position wrist splint as standard conservative care.

Two intervention groups will additionally receive either neurodynamic mobilization exercises or carpal bone mobilization techniques administered by a physiotherapist for four weeks. Clinical outcomes and median nerve morphology will be evaluated at baseline and immediately after the intervention period.

The primary outcome is the change in the Boston Carpal Tunnel Questionnaire score. Secondary outcomes include pain intensity, neuropathic pain, functional disability, muscle strength, pressure pain threshold, and ultrasonographic measurements of the median nerve.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild-to-moderate carpal tunnel syndrome confirmed by electrodiagnostic testing
* CTS symptoms for at least 3 months
* Ability to provide informed consent

Exclusion Criteria:

* Previous carpal tunnel surgery
* Diabetes mellitus or polyneuropathy
* Cervical radiculopathy
* Pregnancy or breastfeeding
* Central nervous system disorders

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire (BCTQ) Total Score | Baseline to 4 weeks
  Change in Boston Carpal Tunnel Questionnaire (BCTQ) Total Score

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline to 4 weeks
  Pain intensity measured using a 10-cm visual analog scale.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | Baseline to 4 weeks
  Change in Neuropathic Pain Score Assessed by Leeds Assessment of Neuropathic Symptoms and Signs (LANSS).
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | Baseline to 4 weeks
  Change in Upper Extremity Disability Assessed by Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH).
Grip Strength | Baseline to 4 weeks
  Change Grip strength measured using a Jamar dynamometer.
Pinch Strength | Baseline to 4 weeks
  Change in Pinch Strength measured using a Pinchmeter.
Pressure Pain Threshold | Baseline to 4 weeks
  Change in pressure pain threshold assessed using J -Tech algometer.
Median Nerve Cross-Sectional Area | Baseline to 4 weeks
  Change in Median Nerve Cross-Sectional Area Assessed by Ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akdeniz Leblebicier, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University Yoncalı Physical Therapy and Rehabilitation Hospital, Kütahya, Yoncalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No